CLINICAL TRIAL: NCT01958957
Title: A Multicenter Safety Clinical Trial of Ginkgolides Meglumine Injection in the Treatment of Ischemic Stroke With Syndrome of Intermingled Phlegm and Blood Stasis.
Brief Title: A Safety Study of Ginkgolides Meglumine Injection in the Treatment of Ischemic Stroke.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201311BDY04V05
Record Dates: First submitted 2013-09-29; First posted 2013-10-09 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2013-05

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; safety; Ginkgolides Meglumine Injection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ginkgolides Meglumine Injection (Experimental): Intravenous drip slowly. A 1 (25 mg), will be taken slowly into the 0.9% sodium chloride injection diluted in 250 ml before use, then slow intravenous drip, once a day. The dripping speed must be strictly controlled. For the first time when using, dripping speed should be controlled for 10 ~ 15 drops per minute. After 30 minutes treatment without discomfort, dripping speed can be appropriately increased, but no more than 30 drops per minute.
  Interventions: Drug: Ginkgolides Meglumine Injection

INTERVENTIONS:
Drug: Ginkgolides Meglumine Injection — 25mg, intravenous drip, once a day. Number of Cycles: 14 days.

SUMMARY:
The aim of this study is to evaluate the safety of Ginkgolides Meglumine Injection in the treatment of ischemic stroke with Syndrome of Intermingled Phlegm and Blood Stasis.

DETAILED DESCRIPTION:
Ginkgolides Meglumine Injection was jointly developed by China Pharmaceutical University and Jiangsu Kanion Pharmaceutical Co., Ltd. Its pharmacal ingredients are ginkgo lactones , ginkgo lactone B, ginkgo lactone K, etc; Excipients for meglumine, citric acid, sodium chloride. It is used to treat stroke (mild-to-moderate cerebral infarction) in recovery phlegm and Syndrome of Intermingled Phlegm and Blood Stasis.

The aim of this study is to evaluate the safety of Ginkgolides Meglumine Injection in the treatment of ischemic stroke with Syndrome of Intermingled Phlegm and Blood Stasis.

ELIGIBILITY:
Inclusion Criteria:

* patients according to diagnostic standards on western medical ischemic stroke;
* patients according to diagnostic standards on Chinese medical attack to meridians;
* patients according to differentiation standards on syndrome of intermingled phlegm and blood stasis;
* 2 weeks to 6 months after attack;
* Age between 18-80 years;
* patients must volunteer to participate in this study and sign the informed consent form.

Exclusion Criteria:

* patients accompanying unconsciousness or severe dementia;
* ALT, AST≥2 times of upper limit of normal;
* patients with other severe diseases such as disease in circulatory system, hematopoietic system, digestive system, endocrine system etc;
* patients allergic to Ginkgo biloba drugs，Meglumine and meglumine agents;
* patients who are pregnant, lactating or planning for pregnancy;
* patients with insanity;
* patients who are not suitable for clinical trial under doctors' consideration;
* patients with Merge bleeding after infarction or patients with hemorrhagic tendency;
* patients with lower extremity venous thrombosis;
* patients who have participated in other clinical trial within 1 month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6300 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 14 days

SECONDARY OUTCOMES:
vital signs after 10 minutes of stasis. | 0，14 days
Blood routine tests | 0, 14 days
ECG | 0, 14 days
Patient- reported outcomes,PRO | 0, 14 days
liver function tests | 0, 14 days
kidney function tests | 0, 14 days
urine routine tests | 0, 14 days
stool routine +occult blood tests | 0, 14 days
Coagulation function tests | 0, 14 days

OTHER OUTCOMES:
NIH Stroke Scale，NIHSS | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gao Ying, Doctor, Principal Investigator — Dongzhimen Hospital, Beijing; Zhou Li, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (86):
- China (86):
  - CN051, Anyang
  - CN071, Baoding
  - CN072, Baoding
  - CN073, Baoding
  - CN027, Baotou
  - CN054, Baotou
  - CN001, Beijing
  - CN083, Beijing
  - CN050, Binzhou
  - CN080, Cangzhou
  - CN041, Changchun
  - CN043, Changchun
  - CN029, Changzhi
  - CN079, Chenzhou
  - CN007, Dalian
  - CN044, Daqing
  - CN018, Daqing
  - CN078, Handan
  - CN063, Ha’erbin
  - CN045, Ha’erbin
  - CN059, Ha’erbin
  - CN046, Ha’erbin
  - CN076, Ha’erbin
  - CN035, Hefei
  - CN036, Hefei
  - CN024, Hegang
  - CN025, Hegang
  - CN042, Hegang
  - CN052, Hengshui
  - CN002, Hengyang
  - CN026, Hohhot
  - CN070, Huaihua
  - CN084, Huaihua
  - CN077, Huanggang
  - CN040, Jiamusi
  - CN062, Jilin
  - CN022, Jilin
  - CN058, Jilin
  - CN030, Jinan
  - CN021, Jingdezhen
  - CN057, Jinzhou
  - CN075, Jiujiang
  - CN088, Jiujiang
  - CN069, Ji’an
  - CN085, Ji’an
  - CN014, Kaifeng
  - CN055, Lianyungang
  - CN013, Luohe
  - CN087, Luoyang
  - CN074, Luoyang
  - CN056, Mudanjiang
  - CN060, Mudanjiang
  - CN061, Mudanjiang
  - CN068, Nanchang
  - CN003, Nanjing
  - CN049, Sanming
  - CN048, Shenyang
  - CN008, Shenyang
  - CN006, Shenyang
  - CN017, Shenyang
  - CN005, Shenzhen
  - CN023, Siping
  - CN016, Suihua
  - CN028, Taiyuan
  - CN020, Tangshan
  - CN019, Tangshan
  - CN034, Tianjin
  - CN033, Tianjin
  - CN082, Wuhan
  - CN032, Wuhan
  - CN012, Xi'an
  - CN010, Xi'an
  - CN031, Xianning
  - CN011, Xianyang
  - CN009, Xianyang
  - CN064, Xinyu
  - CN065, Xinyu
  - CN004, Yancheng
  - CN066, Yichun
  - CN067, Yichun
  - CN047, Yiyang
  - CN038, Yuncheng
  - CN039, Zhenjiang
  - CN015, Zhumadian
  - CN081, Zhuozhou
  - CN053, Zibo